CLINICAL TRIAL: NCT02207647
Title: Prevalence of Pathogens in Cerebrospinal Fluid Obtained From Emergency Department Patients
Status: Terminated | Type: Observational
Why Stopped: Funding used up
Sponsor: Olive View-UCLA Education & Research Institute (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, David A. Talan, Principal Investigator, Olive View-UCLA Education & Research Institute
Other Study IDs: 12H-770352; U01CK000176 (NIH)
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Meningoencephalitis; Other Syndromes Requiring Lumbar Puncture in Emergency Department
MeSH Terms: conditions — Meningoencephalitis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cerebrospinal fluid and blood serum are being collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with syndromes requiring lumbar puncture
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
Of all emergency room patients, persons presenting with encephalitis/meningitis syndrome of a potentially infectious nature are among those of greatest concern. Routine clinical and laboratory evaluation of such patients involves screening for known infectious disease agents, selection of which is nonstandardized. Progress in diagnostic technologies, especially molecular techniques based on genetic characteristics of potential pathogens, has greatly expanded the investigators capacity to evaluate specimens from patients for a much wider range of potential pathogens (bacterial, viral, fungal and parasitic agents). Use of Polymerase Chain Reaction (PCR) technology offers the possibility of identifying causative agents for the approximately 50% of all such presentations which go un-diagnosed. The investigators propose a study involving a collaboration between the EMERGEncy ID NET, a network of 10 geographically diverse university-affiliated urban emergency departments (coordinated by Olive View-UCLA Medical Center) and the Centers for Disease Control and Prevention (CDC), to use these new technologies to address this issue.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 3 months old
* Receiving a Lumbar Puncture in the emergency department as part of their standard care.

Exclusion Criteria:

* No CSF available

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will be conducted by the Emergency ID Net Study group (P.I. David Talan), which consists of a network of 10 emergency departments in university-affiliated hospitals throughout the United States.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2014-04; Primary Completion 2016-07 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
prevalence of pathogens | 2 years
  We will describe the range and proportion of pathogens found in CSF among patients enrolled over a 2 year period.

CONTACTS AND LOCATIONS:
Locations (1):
- Olive View-UCLA Medical Center, Sylmar, California, United States